CLINICAL TRIAL: NCT05830695
Title: Clinical, Radiographic and Tomographic Evaluation of Apexogenesis With Human Treated Dentin Matrix in Young Permanent Molars
Brief Title: Evaluation of Apexogenesis With Human Treated Dentin Matrix in Young Permanent Molars
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: nora mostafa mohammed abo shanady (Other)
Responsible Party: Sponsor-Investigator, nora mostafa mohammed abo shanady, Assistant lecturer at pediatric dentistry oral health and preventive dentistry department, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-3456
Record Dates: First submitted 2023-03-31; First posted 2023-04-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Dentin Bridge
MeSH Terms: interventions — mineral trioxide aggregate; Pemetrexed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human treated dentin matrix (Experimental): study group
  Interventions: Drug: human treated dentin matrix
- mineral tri oxide aggregate (Experimental): control group
  Interventions: Drug: Mineral Trioxide Aggregate

INTERVENTIONS:
Drug: human treated dentin matrix — human treated dentin matrix is compared with mineral trioxide aggregate in apexogenesis
  Other Names: human partially demineralized treated dentin matrix
  Arms: human treated dentin matrix
Drug: Mineral Trioxide Aggregate — mineral trioxide aggregate was used as control
  Other Names: MTA
  Arms: mineral tri oxide aggregate

SUMMARY:
Assess the clinical, radiographic, and tomographic outcomes of apexogenesis with human treated dentin matrix in young permanent molars compared to MTA.

DETAILED DESCRIPTION:
The study was conducted as a split-mouth randomized clinical trial, approved by research ethics committee, Faculty of Dentistry, Tanta University, and carried out at Pediatric Dentistry Department, Faculty of Dentistry, Tanta University. The material preparation was conducted at Pharmaceutical Technology Department, Faculty of Pharmacy, Tanta University. 20 children of both sexes aged from 6 to 8 years old were selected with bilateral deeply carious young permanent mandibular first molars that are indicated for vital pulp therapy.The selected deeply carious molars were randomly divided into two groups as follows:

Group I (Study group): 20 molars were treated with human TDM. Group II: (Control group): 20 molars were treated with White MTA. The participating cases were evaluated clinically and radiographically after 6, 12 and 18 months. Tomographic evaluation was performed immediate postoperatively and at 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral immature permanent mandibular first molars with deep carious lesions.
2. Positive response to pulp testing.
3. Normal radiographic appearance.
4. Healthy children without any systemic disease that interferes with pulp healing.
5. Patient and parent cooperation.

Exclusion Criteria:

1. Clinical signs and symptoms of irreversible pulpitis as spontaneous throbbing pain, tenderness to percussion, abnormal tooth mobility, swelling, or sinus tract.
2. Presence of periapical lesion, external or internal root resorption.
3. Carious furcation involvement.
4. Dystrophic calcification of the pulp.
5. Non restorable tooth.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
clinical outcome | 18 months
  patient reported pain or tenderness on palpation or percussion
clinical outcome | 18 months
  patient/ clinician observed swelling or sinus tract observation
clinical outcome | 18 months
  tooth mobility clinically assessed by grades
radiographic outcomes | 18 months
  radicular changes assessed by clinician from digital periapical radiograph
radiographic outcomes | 18 months
  interradicular changes assessed by clinician from digital periapical radiograph
radiographic outcomes | 18 months
  peri-radicular changes assessed by clinician from digital periapical radiograph
tomographic evaluation | 18 months
  evidence of continuity of root development measured from cone beam computed tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li R, Guo W, Yang B, Guo L, Sheng L, Chen G, Li Y, Zou Q, Xie D, An X, Chen Y, Tian W. Human treated dentin matrix as a natural scaffold for complete human dentin tissue regeneration. Biomaterials. 2011 Jul;32(20):4525-38. doi: 10.1016/j.biomaterials.2011.03.008. Epub 2011 Mar 31. PMID 21458067
- [Background] Tabatabaei FS, Tatari S, Samadi R, Torshabi M. Surface characterization and biological properties of regular dentin, demineralized dentin, and deproteinized dentin. J Mater Sci Mater Med. 2016 Nov;27(11):164. doi: 10.1007/s10856-016-5780-8. Epub 2016 Sep 21. PMID 27655430
- [Background] Widbiller M, Eidt A, Wolflick M, Lindner SR, Schweikl H, Hiller KA, Buchalla W, Galler KM. Interactive effects of LPS and dentine matrix proteins on human dental pulp stem cells. Int Endod J. 2018 Aug;51(8):877-888. doi: 10.1111/iej.12897. Epub 2018 Feb 17. PMID 29377169
- [Background] Chen J, Cui C, Qiao X, Yang B, Yu M, Guo W, Tian W. Treated dentin matrix paste as a novel pulp capping agent for dentin regeneration. J Tissue Eng Regen Med. 2017 Dec;11(12):3428-3436. doi: 10.1002/term.2256. Epub 2017 Feb 15. PMID 28198096
- [Background] Mehrvarzfar P, Abbott PV, Mashhadiabbas F, Vatanpour M, Tour Savadkouhi S. Clinical and histological responses of human dental pulp to MTA and combined MTA/treated dentin matrix in partial pulpotomy. Aust Endod J. 2018 Apr;44(1):46-53. doi: 10.1111/aej.12217. Epub 2017 Aug 18. PMID 28833942